CLINICAL TRIAL: NCT03223558
Title: Early Initiation of Cardiac Rehabilitation Exercise Training After Sternotomy: A Randomised Controlled Trial and Economic Evaluation
Brief Title: Early Initiation of Post Sternotomy CArdiac Rehabilitation
Acronym: SCAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Collaborators: Coventry University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SE191516
Record Dates: First submitted 2017-07-05; First posted 2017-07-21 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Coronary Artery Disease; Aortic Valve Disease; Mitral Valve Disease
Keywords: cardiac rehabilitation
MeSH Terms: conditions — Coronary Artery Disease; Aortic Valve Disease

STUDY DESIGN:
Intervention Model Description: A single blinded parallel group randomised controlled trial will be used to determine non-inferiority of early (2 weeks post operation) vs usual care (6 weeks post operation ) CR for a period of 8 weeks.
Who Masked: Outcomes Assessor
Masking Description: researchers will be blinded during baseline assessment prior to group allocation.
  Participants and the clinical CR team will know the group allocation and therefore cannot be blinded. University hospitals for Coventry and Warwickshire NHS trust research and design department will generate the randomisation sequence remotely using permuted block randomisation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early rehab group (Experimental): start of 8 weeks cardiac rehabilitation 2 weeks following surgery
  Interventions: Behavioral: timing of initiation of cardiac rehabilitation
- usual care group (Active Comparator): start 8 weeks of cardiac rehabilitation 6 weeks post surgery
  Interventions: Behavioral: timing of initiation of cardiac rehabilitation

INTERVENTIONS:
Behavioral: timing of initiation of cardiac rehabilitation — earlier timing of cardiac rehabilitation

SUMMARY:
The main objective of this trial is to investigate the effects of starting exercise rehabilitation earlier than current practice after coronary artery bypass graft(CABG) or Aortic/Mitral valve replacement (VR) surgery.

DETAILED DESCRIPTION:
The trial will compare health improvements after cardiac rehabilitation, (CR) between participants randomly allocated to one of two groups: an early CR group starting exercise after 2 weeks, and a usual care group starting at 6 weeks. It will also collect information on the financial cost of earlier CR to both the health service and the patients.

All primary and secondary outcome measures will be taken at baseline (1 week) and repeated at the start and end of 8 weeks exercise rehabilitation program (2 and 10 weeks from baseline for the early group, 6 and 14 weeks in the usual care group respectively) and at 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery bypass graft, and mitral/aortic valve replacement patients recovering from sternotomy procedure eligible for cardiac rehabilitation
* Able to provide written informed consent
* Male or female 18 years of age or greater

Exclusion Criteria:

* Patients with any of the following:

  * Serious cardiac arrhythmias
  * Current neurological disorders or previous Cerebral Vascular Accident with residual neurological deficit significant enough to limit exercise
  * Enrolled on another clinical trial that involved exercise
  * Unable to enroll for duration of study
* Patients who are unable to provide written consent.
* Patients under the age of 18 or over the age of 90.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2020-08-05 (Actual)

PRIMARY OUTCOMES:
Change in Six Minute Walk Test Distance | Early Group- Change between baseline, 2 weeks post-surgery, 10 weeks post-surgery, and 12-month follow-up. Usual care group- Change between baseline, 6 weeks post-surgery and 14 weeks post-surgery and 12 months follow-up.
  Distance walked unassisted in 6 minutes

SECONDARY OUTCOMES:
Five Times Sit to Stand (Timed) | Early Group- Change between baseline, 2 weeks post-surgery, 10 weeks post-surgery, and 12-month follow-up. Usual care group- Change between baseline, 6 weeks post-surgery and 14 weeks post-surgery and 12 months follow-up.
  Time taken to stand up and sit down five times
Handgrip Strength | Early Group- Change between baseline, 2 weeks post-surgery, 10 weeks post-surgery, and 12-month follow-up. Usual care group- Change between baseline, 6 weeks post-surgery and 14 weeks post-surgery and 12 months follow-up.
  Participant squeezes dynamometer as forcefully as possible. 3 times in each hand.
Leg Strength | Early Group- Change between baseline, 2 weeks post-surgery, 10 weeks post-surgery, and 12-month follow-up. Usual care group- Change between baseline, 6 weeks post-surgery and 14 weeks post-surgery and 12 months follow-up.
  Isometric quadriceps extension. Measured using a dynamometer.
Euroqol 5 Dimensions Questionnaire | Early Group- Change between baseline, 2 weeks post-surgery, 10 weeks post-surgery, and 12-month follow-up. Usual care group- Change between baseline, 6 weeks post-surgery and 14 weeks post-surgery and 12 months follow-up.
  Quality of life/cost benefit analysis questionnaire
Short Form (SF) -12 Questionnaire | Early Group- Change between baseline, 2 weeks post-surgery, 10 weeks post-surgery, and 12-month follow-up. Usual care group- Change between baseline, 6 weeks post-surgery and 14 weeks post-surgery and 12 months follow-up.
  12 Question Quality of Life Questionnaire
Combined General Anxiety Disorder (GAD)-7 and Patient Health Questionnaire(PHQ) 9 | Early Group- Change between baseline, 2 weeks post-surgery, 10 weeks post-surgery, and 12-month follow-up. Usual care group- Change between baseline, 6 weeks post-surgery and 14 weeks post-surgery and 12 months follow-up.
  General Anxiety and Depression Questionnaire
Client Service Receipt Inventory (CSRI) Questionnaire | Early Group- Change between baseline, 10 weeks post-surgery, and 12-month follow-up. Usual care group- Change between baseline, 14 weeks post-surgery and 12 months follow-up
  health service use questionnaire for economic analysis

OTHER OUTCOMES:
Adverse Events | 12 months from surgery.
  Number, type and severity of adverse events during trial

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A Ennis, Principal Investigator — UHCW NHS trust
Locations (1):
- UHCW NHS trust, Coventry, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ennis S, Lobley G, Worrall S, Evans B, Kimani PK, Khan A, Powell R, Banerjee P, Barker T, McGregor G. Effectiveness and Safety of Early Initiation of Poststernotomy Cardiac Rehabilitation Exercise Training: The SCAR Randomized Clinical Trial. JAMA Cardiol. 2022 Aug 1;7(8):817-824. doi: 10.1001/jamacardio.2022.1651. PMID 35731506
- [Derived] Ennis S, Lobley G, Worrall S, Powell R, Kimani PK, Khan AJ, Banerjee P, Barker T, McGregor G. Early initiation of post-sternotomy cardiac rehabilitation exercise training (SCAR): study protocol for a randomised controlled trial and economic evaluation. BMJ Open. 2018 Mar 23;8(3):e019748. doi: 10.1136/bmjopen-2017-019748. PMID 29574443